CLINICAL TRIAL: NCT03821051
Title: China Structural Ventricular Arrhythmias Registry, a Multicenter，Observational and Prospective Study.
Brief Title: China Structural Ventricular Arrhythmias Registry
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Renmin Hospital of Wuhan University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Second Affiliated Hospital of Nanchang University (Other); Sir Run Run Shaw Hospital (Other); West China Hospital (Other); Beijing Anzhen Hospital (Other); General Hospital of Shenyang Military Region (Other); Xuzhou Central Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-950-1
Record Dates: First submitted 2019-01-27; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2018-10

CONDITIONS: Ventricular Arrythmia
Keywords: structural ventricular arrythmia; ischemic cardiomyopathy; arrhythmogenic right ventricular cardiomyopathy; dilated cardiomyopathy; hypertrophic cardiomyopathy; risk stratification
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia; Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — blood sample will be collected from enrolled participants to detect biomarkers, like genes, inflammatory factors ,etc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, prospective, multi-center registry ,aiming at building a risk stratification for malignant structural ventricular arrhythmias. 2000 participants will be recruited from 10 centers in China,with clinical data to be abstracted from medical records ,and blood samples to be collected for finding promising risk indicators.The follow-up should be made every 6 mouths.

DETAILED DESCRIPTION:
In China, the prevalence and risk factors of malignant ventricular arrhythmias remain unclear. In addition ,the mainstream treatment relies on implantable devices and medication.China Malignant Ventricular Arrhythmias Study is a nation-wide complex consisting of several interrelated studies, with the aim of building a risk stratification as well as a efficient and economic strategy for early prevention and treatment.

Structural Ventricular Arrhythmias Registry, as a part of China Malignant Ventricular Arrhythmias Study, is an observational, prospective, multi-center registry, aiming at building a risk stratification for malignant structural ventricular arrhythmias. 2000 patients with definitive diagnosis will be recruited consecutively from 10 major arrhythmia centers distributed in 6 areas in China. At study entry, participants will be interviewed and asked to sign the informed consent. Demographic characteristics, medical history, clinical features, laboratory tests, imaging pictures, medications, procedures, and in-hospital outcomes of patients will be abstracted from medical records by well trained staffs .At the same time, blood samples will be collected to detect biological markers, like genes, inflammatory factors ,etc. Once enrolled, the participants will receive follow up every 6 mouths about condition of arrhythmia, medication, clinical events, etc.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as ventricular arrhythmia resulted by structural heart diseases, including ischemic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, dilated cardiomyopathy, hypertrophic cardiomyopathy, etc.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In 10 major arrhythmia centers distributed in 6 areas in China, 2000 patients satisfying the inclusion criteria will be enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-10-24 (Actual); Primary Completion 2022-10-24 (Estimated); Study Completion 2027-10-24 (Estimated)

PRIMARY OUTCOMES:
sustained tachycardia/ ventricular fibrillation or sudden cardiac death | 5 years
  event of sustained ventricular tachycardia/ ventricular fibrillation or sudden cardiac death

SECONDARY OUTCOMES:
episodes of arrhythmia | 5 years
  record: type of arrhythmia, the amount of episodes, duration, unstable hemodynamics，treatment，
all-cause death | 5 years
  exclude accidents, like trauma, drowning.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Yao, MD,PhD, Study Chair — China National Center for Cardiovascular Diseases
Locations (1):
- China National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China